CLINICAL TRIAL: NCT00255047
Title: Comparative Immunogenicity of Different Multivalent Component Pertussis Vaccine Formulations Based on a 5 Component Acellular Pertussis Vaccine in Infants and Toddlers
Brief Title: Safety and Immune Response of Different Pediatric Combination Vaccines.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M5A10
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2010-11-10 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Diphtheria; Polio; Pertussis
Keywords: Pertussis; Whooping cough; Filamentous Haemagglutinin; Fimbriae Types 2 and 3;; Pertactin; Diphtheria; Tetanus; Poliovirus Types 1, 2, and 3.
MeSH Terms: conditions — Diphtheria; Poliomyelitis; Whooping Cough; Tetanus | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Poliovirus Vaccine, Inactivated; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; pentacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Study Group 1: DAPTACEL®, ActHIB®, and IPOL® (Experimental): Participants will receive 3 doses of DAPTACEL®, ActHIB®, and IPOL® at Months 2, 4, and 6, respectively
  Interventions: Biological: DAPTACEL®. (DTaP), IPOL®., and ActHIB®.
- Study Group 2: Pentacel® (Experimental): Participants will receive 3 doses of Pentacel® at Months 2, 4, and 6, respectively
  Interventions: Biological: Pentacel®: DTaP-IPV/Hib combined
- Study Group 3: DTaP-IPV and ActHIB® (Experimental): Participants will receive 3 doses of DTaP-IPV and ActHIB® at Months 2, 4, and 6, respectively
  Interventions: Biological: DTaP-IPV and ActHIB®
- Study Group 4: Pentacel® (Experimental): Participants will receive 3 doses of Pentacel® at Months 2, 4, and 6, respectively
  Interventions: Biological: Pentacel®: DTaP-IPV/Hib combined

INTERVENTIONS:
Biological: DAPTACEL®. (DTaP), IPOL®., and ActHIB®. — 0.5 mL, Intramuscular
  Other Names: DAPTACEL®; IPOL®; ActHIB®
  Arms: Study Group 1: DAPTACEL®, ActHIB®, and IPOL®
Biological: Pentacel®: DTaP-IPV/Hib combined — 0.5 mL, Intramuscular
  Other Names: Pentacel®
  Arms: Study Group 2: Pentacel®
Biological: DTaP-IPV and ActHIB® — 0.5 mL, Intramuscular
  Other Names: ActHIB®
  Arms: Study Group 3: DTaP-IPV and ActHIB®
Biological: Pentacel®: DTaP-IPV/Hib combined — 0.5 mL, Intramuscular
  Other Names: Pentacel®
  Arms: Study Group 4: Pentacel®

SUMMARY:
The overall aim of the study is to corroborate that a schedule consisting of 3 doses of Pentacel™ and a 4th dose of DAPTACEL® and ActHIB® or 4 doses of Pentacel™ or 4 doses of Quadracel and ActHIB® is as safe and immunogenic as a standard of care schedule based on 3 doses of the licensed-equivalent vaccines DAPTACEL®, Vero cell derived Inactivated Poliovirus vaccine (IPOL®), and ActHIB® and a 4th dose of DAPTACEL® and ActHIB®.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 42 days and ≤ 89 days on the day of inclusion
* Born at full term of pregnancy (≥ 36 weeks)
* Informed consent form signed by the parent(s) or other legally authorized representative(s) before the 1st study related procedure
* Vaccination with a hepatitis B vaccine at least 30 days before inclusion
* Able to attend all scheduled visits and to comply with all trial procedures(i.e., access to a phone)
* Provide blood sample prior to Dose 1
* Parent or legal representative willing to take rectal temperatures after each vaccination.

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the (first)trial vaccination
* Planned participation in another clinical trial during the present trial period
* Personal or immediate family history of congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Known or suspected systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing the same substances as the trial vaccine(s)
* Chronic illness that could interfere with trial conduct or completion
* Received blood or blood-derived products since birth
* Any vaccination in the 2 weeks preceding the first trial vaccination or planned in the 4 weeks after any trial vaccination. Flu vaccine could be administered only 2 weeks after any trial vaccination
* Previous vaccination with any acellular pertussis- (DTaP) or whole cell pertussis- (DTwP) based combination vaccines, Haemophilus influenzae type b (Hib)-conjugate, poliovirus, or pneumococcal conjugate vaccines
* Coagulation disorder contraindicating intramuscular (IM) vaccination
* Clinically significant findings on review of systems (determined by investigator or sub-investigator to be sufficient for exclusion)
* Developmental delay or neurological disorder
* Any condition which, in the opinion of the investigator, would interfere with the evaluation of the vaccine or pose a health risk to the subject.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2167 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (32):
- United States (32):
  - Tuscaloosa, Alabama
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Oakland, California
  - Paramount, California
  - Norwich, Connecticut
  - Palm Beach Gardens, Florida
  - Marietta, Georgia
  - Bardstown, Kentucky
  - Bossier City, Louisiana
  - Baltimore, Maryland
  - Woburn, Massachusetts
  - Omaha, Nebraska
  - Ithaca, New York
  - Liverpool, New York
  - Huber Heights, Ohio
  - Youngstown, Ohio
  - Norristown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Kingsport, Tennessee
  - Amarillo, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Provo, Utah
  - South Jordan, Utah
  - St. George, Utah
  - Spokane, Washington
  - Vancouver, Washington
  - Huntington, West Virginia
  - Marshfield, Wisconsin

REFERENCES:
- [Derived] Chatterjee A, O'Keefe C, Varman M, Klein NP, Luber S, Tomovici A, Noriega F. Comparative immunogenicity and safety of different multivalent component pertussis vaccine formulations and a 5-component acellular pertussis vaccine in infants and toddlers: a randomized, controlled, open-label, multicenter study. Vaccine. 2012 May 14;30(23):3360-8. doi: 10.1016/j.vaccine.2012.03.057. Epub 2012 Apr 1. PMID 22475857
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 10 November 2005 through 21 September 2006 in 38 Clinics in the Untied States.
Pre-assignment Details: A total of 2167 participants that met the inclusion and exclusion criteria were enrolled and vaccinated. Data on Stage I, up to the 3rd dose are presented.
Groups:
- Study Group 1: DAPTACEL®, IPOL®, and ActHIB®: Participants received 3 doses (0.5 mL each) of DAPTACEL®, IPOL®, and ActHIB® at Months 2, 4, and 6, respectively.
- Study Group 2: Pentacel®; Study Group 4: Pentacel®: Participants received 3 doses (0.5 mL each) of Pentacel® at Months 2, 4, and 6 respectively.
- Study Group 3: DTaP-IPV and ActHIB®: Participants received 3 doses (0.5 mL each) of DTaP-IPV and ActHIB® at Months 2, 4, and 6, respectively.
Period: Overall Study
Arm/Group | Study Group 1: DAPTACEL®, IPOL®, and ActHIB® | Study Group 2: Pentacel® | Study Group 3: DTaP-IPV and ActHIB® | Study Group 4: Pentacel®
Started | 538 | 535 | 546 | 548
Completed | 490 | 487 | 496 | 502
Not Completed | 48 | 48 | 50 | 46
Not completed — Serious Adverse Events | 2 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 3 | 2 | 1
Not completed — Protocol Violation | 13 | 13 | 16 | 20
Not completed — Lost to Follow-up | 9 | 8 | 5 | 6
Not completed — Withdrawal by Subject | 24 | 23 | 25 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group 1: DAPTACEL®, IPOL®, and ActHIB® | Study Group 2: Pentacel® | Study Group 3: DTaP-IPV and ActHIB® | Study Group 4: Pentacel® | Total
Number analyzed (Participants) | 538 | 535 | 546 | 548 | 2167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 538 | 535 | 546 | 548 | 2167
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.2 (0.27) | 2.1 (0.27) | 2.2 (0.27) | 2.1 (0.28) | 2.1 (0.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 242 | 249 | 274 | 1016
  Male | 287 | 293 | 297 | 274 | 1151
Region of Enrollment [Number; unit: participants]
  United States | 538 | 535 | 546 | 548 | 2167

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participant Responding to Pertussis Antigens Post-Dose 3 of Pentacel® or DAPTACEL®, IPOL®, and ActHIB® Vaccinations.
Description: Vaccine response was calculated as a pre-dose 1 titer ≤ Lower Limit of Quantitation (LLOQ) and post-dose 3 titer > LLOQ; or a pre-dose 1 titer > LLOQ and post-dose 3 titer ≥ pre-dose 1 titer.
Time Frame: 30 Days post-dose 3 vaccination
Population: The vaccine response to pertussis antigens were determined in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group 1: DAPTACEL®, IPOL®, and ActHIB® | Study Group 2: Pentacel® | Study Group 3: DTaP-IPV and ActHIB® | Study Group 4: Pentacel®
Number analyzed (Participants) | 419 | 405 | 411 | 424
Percentage of Participants
  Pertussis Toxoid (PT) | 98 | 99 | 99 | 99
  Filamentous Haemagglutinin (FHA) | 86 | 96 | 95 | 96
  Pertactin (PRN) | 94 | 92 | 94 | 92
  Fimbriae Types 2 and 3 (FIM) | 97 | 96 | 99 | 97

2. Primary Outcome: Percentage of Participants With a Four-fold Rise in Pertussis Antigens Post-Dose 3 of Pentacel® or DAPTACEL®, IPOL®, and ActHIB® Vaccinations (Seroconversion)
Time Frame: 30 Days post-dose 3 vaccination
Population: Four-fold rise titers (seroconversion) were evaluated in the per-protocol population
Measure: Number; unit: Percentage of participants
Arm/Group | Study Group 1: DAPTACEL®, IPOL®, and ActHIB® | Study Group 2: Pentacel® | Study Group 3: DTaP-IPV and ActHIB® | Study Group 4: Pentacel®
Number analyzed (Participants) | 419 | 405 | 411 | 424
Percentage of participants
  Pertussis Toxoid (PT) | 89 | 92 | 92 | 92
  Filamentous Haemagglutinin (FHA) | 54 | 75 | 77 | 77
  Pertactin (PRN) | 71 | 67 | 76 | 68
  Fimbriae Types 2 and 3 (FIM) | 86 | 85 | 94 | 90

3. Other Pre Specified Outcome: Number of Participants Reporting at Least One Solicited Injection Site or Systemic Reactions Post-vaccination 3
Description: Solicited injection site reactions: Tenderness, Redness, and Swelling. Solicited systemic reactions: Fever (body temperature), Vomiting, Abnormal crying, Lethargy, Appetite decreased, Irritability, and Rash.
Time Frame: 7 days post-vaccination 3
Population: Solicited injection site and systemic reactions were evaluated in the intend-to-treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | Study Group 1: DAPTACEL®, IPOL®, and ActHIB® | Study Group 2: Pentacel® | Study Group 3: DTaP-IPV and ActHIB® | Study Group 4: Pentacel®
Number analyzed (Participants) | 538 | 535 | 546 | 548
Participants
  Any Solicited Injection Site Reaction | 203 | 160 | 164 | 160
  Any Erythema | 34 | 28 | 21 | 18
  Grade 3 Erythema Any dose (>50 mm) | 0 | 1 | 0 | 0
  Any Swelling | 12 | 18 | 10 | 14
  Grade 3 Swelling Any dose (>50 mm) | 0 | 1 | 0 | 0
  Any Tenderness | 186 | 152 | 150 | 148
  Grd 3 Tenderness (cries when inj. limb is moved) | 11 | 4 | 6 | 4
  Any Solicited Systemic Reaction | 311 | 303 | 328 | 309
  Any Fever | 102 | 102 | 124 | 94
  Grade 3 Fever (> 39.5 C) | 3 | 4 | 7 | 1
  Any Vomitting | 49 | 40 | 41 | 42
  Grade 3 Vomitting (≥3 episodes) | 9 | 3 | 3 | 7
  Any Anormal crying | 144 | 114 | 125 | 133
  Grade 3 Abnormal crying (Inconsolable > 3 hrs) | 3 | 1 | 2 | 4
  Any Lethargy | 114 | 97 | 100 | 91
  Grade 3 Lethargy (disabling) | 4 | 0 | 4 | 0
  Any Appetite decreased | 84 | 72 | 85 | 65
  Grade 3 Appetite decreased (skips ≥ 2 meals) | 4 | 0 | 3 | 1
  Any Irritability | 242 | 239 | 254 | 242
  Grade 3 Irritability (continuously for >3 hours) | 5 | 12 | 11 | 11

4. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies to Pentacel® or DAPTACEL®, IPOL®, and ActHIB® Antigens Post-dose 3 Vaccinations.
Time Frame: 30 Days post-dose 3 vaccination.
Population: Geometric mean titers were evaluated in the per-protocol immunogenicity population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1: DAPTACEL®, IPOL®, and ActHIB® | Study Group 2: Pentacel® | Study Group 3: DTaP-IPV and ActHIB® | Study Group 4: Pentacel®
Number analyzed (Participants) | 422 | 406 | 414 | 425
Titers
  Pertussis Toxoid (EU/mL) | 66.48 [62.54 to 70.67] | 96.8 [91.4 to 102.4] | 116.86 [110.60 to 123.47] | 97.8 [92.5 to 103.3]
  Filamentous Haemagglutinin (EU/mL) | 22.51 [20.94 to 24.20] | 53.0 [49.7 to 56.6] | 56.88 [53.26 to 60.74] | 54.1 [50.9 to 57.4]
  Pertactin (EU/mL) | 33.63 [30.92 to 36.58] | 32.5 [29.5 to 35.9] | 44.70 [40.95 to 48.80] | 32.5 [29.5 to 35.8]
  Fimbriae Types 2 and 3 (EU/mL) | 181.66 [166.62 to 198.06] | 188.5 [173.9 to 204.3] | 273.10 [254.83 to 292.67] | 199.0 [184.3 to 214.8]
  Polyribosylribitol Phosphate-Tetanus Toxoid; μg/mL | 2.38 [2.01 to 2.81] | 2.5 [2.2 to 2.9] | 3.76 [3.25 to 4.34] | 2.5 [2.2 to 2.9]
  Diphtheria (IU/mL) | 0.32 [0.29 to 0.36] | 0.3 [0.3 to 0.4] | 0.37 [0.33 to 0.41] | 0.3 [0.3 to 0.3]
  Tetanus toxoid (IU/mL, ≥ 0.01) | 0.97 [0.91 to 1.04] | 0.8 [0.7 to 0.8] | 1.09 [1.02 to 1.17] | 0.8 [0.7 to 0.8]
  Poliovirus Types 1 (≥ 1:8 dil) | 719.83 [645.73 to 802.42] | 397.7 [342.8 to 461.5] | 776.44 [676.85 to 890.68] | 468.3 [406.3 to 539.8]
  Poliovirus Types 2 (≥ 1:8 dil) | 734.50 [668.28 to 807.28] | 699.5 [623.6 to 784.6] | 1203.20 [1082.31 to 1337.60] | 812.5 [727.3 to 907.7]
  Poliovirus Types 3 (≥ 1:8 dil) | 916.90 [829.15 to 1013.92] | 666.6 [584.7 to 760.0] | 1115.00 [976.11 to 1273.65] | 819.9 [715.8 to 939.0]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for 4 months post-vaccination 1 (Stage I)
Arm/Group | Study Group 1: DAPTACEL®, IPOL®, and ActHIB® | Study Group 2: Pentacel® | Study Group 3: DTaP-IPV and ActHIB® | Study Group 4: Pentacel®
Serious Adverse Events (participants affected / at risk) | 18/538 | 18/535 | 21/546 | 11/548
Other Adverse Events (participants affected / at risk) | 399/538 | 394/535 | 421/546 | 414/548
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group 1: DAPTACEL®, IPOL®, and ActHIB® (N=538) | Study Group 2: Pentacel® (N=535) | Study Group 3: DTaP-IPV and ActHIB® (N=546) | Study Group 4: Pentacel® (N=548)
Congenital aortic anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acquired pyloric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper extremity mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 7 (7) | 4 (4) | 6 (6) | 3 (3)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kawasaki´s disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General nutrition disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (3)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotonic-hyporesponsive episode (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Study Group 1: DAPTACEL®, IPOL®, and ActHIB® (N=538) | Study Group 2: Pentacel® (N=535) | Study Group 3: DTaP-IPV and ActHIB® (N=546) | Study Group 4: Pentacel® (N=548)
Diarrhoea (Gastrointestinal disorders) | 39 (44) | 34 (37) | 41 (43) | 41 (43)
Teething (Gastrointestinal disorders) | 35 (44) | 33 (43) | 30 (40) | 34 (48)
Pyrexia (General disorders) | 27 (35) | 33 (34) | 22 (25) | 25 (27)
Bronchiolitis (Infections and infestations) | 24 (27) | 34 (37) | 28 (30) | 16 (17)
Otitis media (Infections and infestations) | 72 (86) | 97 (117) | 93 (109) | 75 (94)
Upper respiratory tract infection (Infections and infestations) | 143 (164) | 141 (167) | 134 (162) | 141 (167)
Viral infection (Infections and infestations) | 16 (17) | 31 (32) | 20 (22) | 23 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (42) | 49 (54) | 45 (51) | 44 (47)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 51 (59) | 49 (57) | 50 (59) | 42 (46)
Injection site erythema (General disorders) | 90/532 (174) | 65/533 (83) | 64/538 (107) | 66/543 (82)
Injection site swelling (General disorders) | 49/532 (102) | 50/533 (59) | 43/538 (77) | 49/543 (71)
Injection site pain (General disorders) | 342/532 (1406) | 310/533 (545) | 301/538 (967) | 310/543 (542)
Fever (General disorders) | 219/531 (300) | 199/533 (254) | 221/537 (304) | 208/543 (268)
Vomiting (Gastrointestinal disorders) | 128/532 (169) | 119/533 (153) | 131/538 (174) | 119/543 (150)
Anbormal crying (Psychiatric disorders) | 287/532 (495) | 282/533 (446) | 275/539 (452) | 285/543 (442)
Lethargy (General disorders) | 271/532 (456) | 275/533 (415) | 262/538 (415) | 239/543 (369)
Appetite Decreased (Metabolism and nutrition disorders) | 214/532 (295) | 191/533 (253) | 192/538 (267) | 174/543 (251)
Irritability (Psychiatric disorders) | 399/532 (820) | 394/533 (795) | 421/539 (820) | 414/543 (800)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.